CLINICAL TRIAL: NCT05256264
Title: Machine-learning Algorithm to Differentiate Intraoperative Ketamine Dosing Based on Electroencephalographic Density Spectrum Array Analysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-09-008BC
Record Dates: First submitted 2022-02-15; First posted 2022-02-25 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Electroencephalographic Density Spectrum Array Analysis; Density Spectrum Array; Ketamine; Multimodal General Anesthesia
Keywords: General anesthesia; Ketamine; Density Spectrum Array; Electroencephalogram; Multimodal General Anesthesia; Machine learning
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: Sevoflurane
- Low dose ketamine group: Sevoflurane + 3µg/kg/min ketamine infusion
  Interventions: Drug: Ketamine
- High dose ketamine group: Sevoflurane + 6µg/kg/min ketamine infusion
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Ketamine infusion at different dose to observe EEG DSA changes
  Other Names: Ketamine Hydrochloride
  Groups: High dose ketamine group; Low dose ketamine group

SUMMARY:
Ketamine is widely used in the setting of multimodal general anesthesia, and the Electroencephalographic density spectral array (DSA) monitoring has been implemented in the practice of anesthesia. The purpose of this study is to investigate the dose-response EEG changes in patients during the perioperative period when ketamine is used. With the application of machine-learning algorithm, we aim to interpret the ketamine dosing precisely and accurately, based on the DSA obtained.

DETAILED DESCRIPTION:
In this single-blinded randomized controlled trial, we enroll 90 patients undergoing major spine surgery, and candidates are divided into 3 groups: A (control group using sevoflurane only), B (sevoflurane + 3µg/kg ketamine infusion), C (sevoflurane + 6µg/kg/min ketamine infusion). Throughout the perioperative period, under standardized perioperative care, each patient will be monitored with EEG DSA. The data obtained will be utilized for machine-learning in the development of a algorithm to interpret the precise dosing of ketamine in respect of its effect on the EEG DSA. This study is also anticipated to boost the development of dose-response algorithm of other agents, promoting the advancement of the concept of "multimodal general anesthesia"

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective spine surgery
2. Aged 20-80 years old

Exclusion Criteria:

1. Pregnancy
2. Presence of major brain disorders: stroke, epilepsy, Parkinson's disease, etc.
3. Any of the following major organ disorders:

   1. Chronic pulmonary disease (Clinically diagnosed severe chronic obstructive pulmonary disease or FEV1/FVC <70% or FEV1 <50%)
   2. Heart failure (NYHA III or IV)
   3. Chronic renal failure (eGFR<60ml/min/1.73m2)
4. Ongoing sepsis or infection
5. Ongoing of history of CNS-acting medications/substances use (e.g.: sedatives, hypnotics, stimulants, etc.)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted for spine surgery under the department of orthopedic surgery at VGHTPE, a tertiary hospital in Taiwan, will be selected.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Ketamine dosing based on EEG DSA | DSA EEG is placed before anesthesia starts, recorded throughout the operative procedure until emergence and patient is extubated. The saved EEG DSA data will be retrieved by the end of the day.
  The DSA is obtained from raw EEG by fast Fourier transformation. By interpreting the DSA, we can obtain the trends and changes of power within different frequencies over time, in respect to different ketamine dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Kun Ting, MD, PhD, Study Chair — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Beitou, Taiwan